CLINICAL TRIAL: NCT03637881
Title: A Pilot Study Investigating Consumer Perspective and Understanding of the Term "Milk"
Brief Title: Cconsumer Perspective and Understanding of the Term "Milk"
Acronym: CMK
Status: Completed | Type: Observational
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB2018-069
Record Dates: First submitted 2018-07-25; First posted 2018-08-20 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Health Behavior
Keywords: Milk; Consumer choice
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Other: Daily or non-daily Consumers

SUMMARY:
The objectives of this study are:

1. To determine the consumption behaviors of dairy and non-dairy milks across a diverse demographic.
2. To determine the purchasing behaviors of dairy and non-dairy milks across a diverse demographic.
3. To determine the variation in medical history and health conditions amongst consumers of dairy milk and non-dairy milk alternatives.
4. To assess the general knowledge and awareness of health associated with dairy milk and non-dairy milk alternatives.

DETAILED DESCRIPTION:
This study is an observational, cross-sectional trial design focused on obtaining information about consumer understanding and perception of the term "milk" and how they affect consumer choice.

A planned sample size of 50 will be enrolled into the study. This study will require one initial screening visit and 1 Study Day. This study will take approximately 2 to 2 ½ hours per subject to complete.

The initial screening visit will provide subject with the informed consent document and determine subject eligibility through anthropometric measurements, vital signs, and completion of an eating habits questionnaire.

If willing and eligible to participate, subjects will be invited to participate in the study for 1 Study Day that participants can choose to continue on to after the Screening visit.

Subject will arrive at the center in fasted for at least 2 hours or longer. During the Study Day, each participant will be asked to participate in two activities. In the first activity, participants will be presented with eight differently-labeled milk cartons, each accompanied by a fixed price label, and asked to answer questions regarding consumption. In the second activity, participants will be presented with the same setup from the first activity, however, the price labels for each product is varied according to real market prices for each product. In this activity, participants will be asked to answer questions regarding purchasing. Following these two activities, participants will then be asked to answer a questionnaire on consumer choice for dairy and non-dairy milk.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent and comply with procedures

Exclusion Criteria:

* Under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Voluntary to participant to this study
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Data collection of consumption behaviors of dairy and non-dairy milks across a diverse demographic via questionnaire | 30 minutes
  Consumption behaviors of dairy and non-dairy milks

SECONDARY OUTCOMES:
Data collection of purchasing behaviors of dairy and non-dairy milks across a diverse demographic via questionnaire | 30 minutes
  Purchasing behaviors of dairy and non-dairy milks
Data collection of variations in medical history and health conditions amongst consumers of dairy milk and non-dairy milk alternatives via questionnaire | 30 minutes
  variation in medical history and health conditions
Data collection of the general knowledge and awareness of health associated with dairy milk and non-dairy milk alternatives via questionnaire | 30 minutes
  the general knowledge and awareness of health

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States